CLINICAL TRIAL: NCT04333901
Title: Assessment of the Home Non-invasive Compliance in Patients With Chronic Obstructive Pulmonary Disease Following the Introduction of Long-term Ventilation. An Observational Study
Brief Title: Compliance of Long-term Home Non-invasive Ventilation for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Vivisol (Other)
Collaborators: Slb Pharma (Other); France Oxygène (Unknown); MBar (Unknown)
Responsible Party: Sponsor
Other Study IDs: VENTIOBS; IDRCB 2019 A01902-55 (Other: French National Health Agency)
Record Dates: First submitted 2020-03-04; First posted 2020-04-03 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: home non-invasive ventilation; compliance; quality of life; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background : Long-term home non-invasive ventilation (NIV) can be proposed as treatment for acute respiratory failure with severe alveolar hypoventilation. The aim of NIV is to correct both daytime and night-time hypoventilation and associated symptoms and to provide the patient with adequate night-time oxygen saturation. The benefits of long-term NIV in the management of chronic obstructive pulmonary disease (COPD) patients in a stable state remain controversial. This highlights the importance of identifying the predictive factors for good compliance to the NIV, defined as a use of more than 4 hours per day.

Aim of the study: The main objective is this observational study is to monitor the home NIV compliance over a period of 1 year under real conditions of treatment in patients with COPD newly initiated onto NIV (with telemonitoring or not) in order to specify the predictive criteria for good compliance. The secondary objectives are to assess the evolution of functional respiratory data, NIV parameters and changes in prescription, occurrence of acute exacerbations of COPD, hospitalizations and death, patient outcomes (quality of life and acceptability of NIV).

Study design: a cohort of 120 patients with COPD newly initiated onto home-NIV (with telemonitoring or not), either in a stable state or following an acute exacerbation will be enrolled in the study and follow-up over 1 year. Data will be collected by lung specialists and home health care provider teams at 1-month post-initiation of NIV, 6 months and 1 year. The study is conduct in France.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who require the initiation of a home-NIV (in case of previous equipment: NIV interrupted for more than 6 months).
* Life expectancy greater than 1 year.
* Patient who has agreed to participate in the observational study after receiving clear information from the investigator and signing the consent form.

Exclusion Criteria:

* NIV indicated for the treatment of chronic respiratory failure other than COPD.
* Patient with overlap syndrome (COPD associated to OSA).
* Patient with limitations who do not allow proper use of the NIV device.
* Simultaneous participation in a health intervention research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of COPD patients who initiate long-term home-NIV.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the global compliance of the home-NIV over 1 year | 1 year
  For each patient, the total number of hours of NIV use divided by the number of days over the period of observation will be calculated.

SECONDARY OUTCOMES:
Evolution of the mean duration of NIV use per day | month 1, month 6, month 12
  The mean number of hours of NIV use per day will be calculated by period of 30 consecutive days at different times over the year of home NIV introduction.
  At each time, the proportion of patients with NIV use ≥ 4 hours per day will be calculated.
Impact of the home-NIV on the medical condition of COPD patients | 1 year
  The number of hospitalizations, COPD exacerbations, deaths will be monitored over 1 year.
Impact of the home-NIV on the dyspnea | At inclusion, month 6, month 12
  The respiratory function will be evaluated with the score of dyspnea assessed using the Modified Medical Research Council (mMRC) scale.
  The score ranges from 0 to 4 points; higher scores mean a high dyspnea.
Impact of the home-NIV on the respiratory function | At inclusion, month 6, month 12
  The pulmonologist will assess the evolution of respiratory function according to good medical practice with the pulmonary functional tests and blood gas analysis, and judge if the prescribed home-NIV treatment is sufficient to normalize the respiratory function or if the treatment must be modified.
Impact of the home-NIV on the health related quality of life of COPD patients | At inclusion, month 6
  the quality of life will be assessed using the COPD-specific health related quality of life questionnaire named VQ11. The questionnaire VQ11 comprises 11 items distributed across three components (functional: 3 items, psychological: 4 items, social: 4 items). The global score ranges from 11 to 55 points; higher scores mean a better quality of life.
Assessment of home-NIV by patients | month 6
  The home-NIV treatment will be assessed by patients using the S3-NIV questionnaire (this short questionnaire comprises 11 items distributed across three NIV-related components : respiratory Symptoms, Sleep quality and NIV-related Side effects. The global score varies between 0 to 10 points; higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Jébrak, MD, Principal Investigator — Bichat Hospital
Locations (8):
- France (8):
  - Pays d'Aix hospital, Aix-en-Provence
  - Cannes hospital, Cannes
  - Henri-Mondor hospital (APHP), Créteil
  - Institut Médical de Sologne Les Pins, Lamotte-Beuvron
  - Le Havre Jacques Monod hospital, Montivilliers
  - Pitié Salpétrière hospital (APHP), Paris
  - Bichat hospital, Paris
  - Saint-Nazaire hospital, Saint-Nazaire